CLINICAL TRIAL: NCT04405713
Title: Assessment of Different Timing for Early Laparoscopic Cholecystectomy in Acute Calcular Cholecystitis (Multicentric Study)
Brief Title: Different Timing for Early Laparoscopic Cholecystectomy in Acute Calcular Cholecystitis
Acronym: ACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, gastrointestinal surgical center, Mansoura University, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: early LC for ACC
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Acute Cholecystitis
Keywords: Early laparoscopic cholecystectomy; postcholecystectomy bile injury; delay laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Intervention Model Description: Patients with ACC were divided into three groups according to the timing of the surgery: from the onset of symptoms within the first 3 days (group 1), between 4 and 7 days (group 2) and beyond 7 days (group 3).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients were divided into three groups according to the timing of the surgery: from the onset of symptoms within the first 3 days (group 1), between 4 and 7 days (group 2) and beyond 7 days (group 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- from the onset of symptoms within the first 3 days (group 1) (Active Comparator): ELC for ACC from the onset of symptoms within the first 3 days (group 1)
  Interventions: Procedure: from the onset of symptoms within the first 3 days
- from the onset of symptoms within the 4-7 days (Active Comparator): ELC for ACC from the onset of symptoms within the4-7 days (group II)
  Interventions: Procedure: : from the onset of symptoms within the 4-7 days
- from the onset of symptoms beyond 7 days (Active Comparator): ELC for ACC from the onset of symptoms beyond 7 days (group III)
  Interventions: Procedure: from the onset of symptoms beyond 7 days

INTERVENTIONS:
Procedure: from the onset of symptoms within the first 3 days — ELC within 3 days of onset of ACC
  Other Names: group 1
  Arms: from the onset of symptoms within the first 3 days (group 1)
Procedure: : from the onset of symptoms within the 4-7 days — ELC 4-7days of onset of ACC
  Other Names: Group II
  Arms: from the onset of symptoms within the 4-7 days
Procedure: from the onset of symptoms beyond 7 days — ELC after 7days of onset of ACC
  Other Names: Group III
  Arms: from the onset of symptoms beyond 7 days

SUMMARY:
The ideal timing for ELC continues to be debatable in patients with acute calculator cholecystitis (ACC). This study was planned to identify the impact of different ELC timing in ACC on surgical outcomes in terms of safety and efficacy

DETAILED DESCRIPTION:
This multicentric analysis involved of successive patients with ACC ELC between April 2018 and March 2020. Patients were divided into three groups according to the timing of the surgery: from the onset of symptoms within the first 3 days (group 1), between 4 and 7 days (group 2), and beyond 7 days (group 3). The primary outcome was the incidence of postoperative complications The secondary outcomes were conversion rate, blood loss, operative times, operational difficulty, the cost-benefit relationship, postoperative stay with each treatment line.

ELIGIBILITY:
Inclusion Criteria:

ACC patients who underwent early LC

Exclusion Criteria:

Pregnancy, Acalculous cholecystitis, CBDS, Ascending cholangitis, Pancreatitis, ASA score 4, Patients scheduled for DLC with failed medical treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative morbidity | 30 DAYS
  the incidence of postoperative morbidity during the 30th day of postoperative procedure

SECONDARY OUTCOMES:
conversion rate | INTRAOPERATIVE
  conversion rate to open cholecystectomy
blood loss | intraoperative
  blood loss
hospital stay | 30 days
  overall hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ayman E Nakeeb, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Mohamed Attea, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
plan to make individual participant data (
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/en/

REFERENCES:
- [Result] El Zanati H, Nassar AHM, Zino S, Katbeh T, Ng HJ, Abdellatif A. Gall Bladder Empyema: Early Cholecystectomy during the Index Admission Improves Outcomes. JSLS. 2020 Apr-Jun;24(2):e2020.00015. doi: 10.4293/JSLS.2020.00015. PMID 32425482
- [Result] Mora-Guzman I, Di Martino M, Gancedo Quintana A, Martin-Perez E. Laparoscopic Cholecystectomy for Acute Cholecystitis: Is the Surgery Still Safe beyond the 7-Day Barrier? J Gastrointest Surg. 2020 Aug;24(8):1827-1832. doi: 10.1007/s11605-019-04335-5. Epub 2019 Aug 6. PMID 31388885
- [Result] Brunee L, Hauters P, Closset J, Fromont G, Puia-Negelescu S; Club Coelio. Assessment of the optimal timing for early laparoscopic cholecystectomy in acute cholecystitis: a prospective study of the Club Coelio. Acta Chir Belg. 2019 Oct;119(5):309-315. doi: 10.1080/00015458.2018.1529344. Epub 2018 Oct 25. PMID 30354853
- [Result] Inoue K, Ueno T, Nishina O, Douchi D, Shima K, Goto S, Takahashi M, Shibata C, Naito H. Optimal timing of cholecystectomy after percutaneous gallbladder drainage for severe cholecystitis. BMC Gastroenterol. 2017 May 31;17(1):71. doi: 10.1186/s12876-017-0631-8. PMID 28569137
- [Result] Onoe S, Kaneoka Y, Maeda A, Takayama Y, Fukami Y. Feasibility of laparoscopic cholecystectomy for acute cholecystitis beyond 72 h of symptom onset. Updates Surg. 2016 Dec;68(4):377-383. doi: 10.1007/s13304-016-0409-5. Epub 2016 Oct 26. PMID 27785732
- [Result] Menahem B, Mulliri A, Fohlen A, Guittet L, Alves A, Lubrano J. Delayed laparoscopic cholecystectomy increases the total hospital stay compared to an early laparoscopic cholecystectomy after acute cholecystitis: an updated meta-analysis of randomized controlled trials. HPB (Oxford). 2015 Oct;17(10):857-62. doi: 10.1111/hpb.12449. Epub 2015 Jul 27. PMID 26218858
- See also: Mansoura university — http://www.mans.edu.eg/en/
- Available data/document: Study Protocol: Ayman El Nakeeb — http://www.mans.edu.eg/en/ — elnakeebayman@yahoo.com